CLINICAL TRIAL: NCT03206593
Title: Fasting Serum Lipids and Glucose Levels in Relation to CVD Outcomes in Patients With Ischemic Heart Failure
Brief Title: Serum Lipids and Glucose Levels in Relation to CVD Outcomes in Patients With Ischemic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Faye Jiang, Dr., Guangdong Provincial People's Hospital
Other Study IDs: No.GDREC2017128H(R1)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Ischemic Heart Failure; Lipids; Fasting Plasma Glucose; Cardiovascular Outcomes; All-cause Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current prospective cohort study is to evaluate the association between fasting lipid profiles (including total cholesterol, low density lipoprotein-cholesterol, high density lipoprotein-cholesterol, triglycerides, apolipoprotein A, apolipoprotein B and lipoprotein(a)) and fasting plasma glucose at admission with cardiovascular disease outcomes (including fatal and non-fatal myocardial infarction, fatal and non-fatal ischemic stroke, re-hospitalization due to heart failure, revascularization by percutaneous coronary intervention or coronary artery bypass grafting, or cardiovascular mortality) and all-cause mortality.in patients with ischemic heart failure and left ventricular ejection fraction < 45 % evaluated by echocardiography during 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria: 1.Diagnosed as coronary artery disease by coronary angiography; 2. Left ventricular ejection fraction < 45% evaluated by echocardiography during index hospitalization.

-

Exclusion Criteria: Coexistent malignant diseases; stage 3 or more of chronic kidney disease; liver dysfunction with ALT or AST higher than 3 times of normal limit range; do not want to participant in current study

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are diagnosed as coronary artery disease by coronary angiography and also have left ventricular ejection fraction < 45% enroll if qualified to our inclusion criteria and exclusion criteria and informed consent will be provided.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular diseases outcomes | 12 months after discharge from index hospitalization
  Fatal or non-fatal myocardial infarction, fatal or non-fatal ischemic stroke, re-hospitalization due to heart failure, revascularization by percutaneous coronary intervention or coronary artery bypass grafting, and cardiovascular mortality

SECONDARY OUTCOMES:
All-cause mortality | 12 months after discharge from index hospitalization
  All-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China